CLINICAL TRIAL: NCT02160639
Title: Evaluating the Impact of Year Long, Augmented Diabetes Self Management Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American Association of Diabetes Educators (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BMS-DSMES-2014
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes self management education; diabetes self management support; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention): usual care includes diabetes self management education
- diabetes self management support (Active Comparator): diabetes self management support in addition to usual care, which includes diabetes self management education
  Interventions: Other: diabetes self management support

INTERVENTIONS:
Other: diabetes self management support — diabetes self management support is telephonic and provided by health investigators
  Arms: diabetes self management support

SUMMARY:
Improving diabetes social support is associated with health improvement benefits. This study is a prospective randomized controlled trial comparing the effects of telephone-based diabetes self-management support (DSMS) compared with usual care, which includes diabetes self-management education (DSME), during a 1-year period. It will determine whether this specific model for providing on-going support to people with diabetes will better enable them to maintain the engagement in self-care behaviors, clinical improvements and diabetes-specific knowledge gained during the course of diabetes self-management education.

DETAILED DESCRIPTION:
Diabetes self management support is telephonic and will be provided by health navigators at a central call center

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Diagnosis of type 2 diabetes mellitus
* HbA1c > 8
* Have not completed a diabetes self management education program in the past year

Exclusion Criteria:

* Current engagement in cancer treatment
* Diagnosis of end-stage renal disease
* Pregnant
* Receiving immunosuppressant therapy following transplant
* Diagnosis of serious mental illness
* Undergoing systemic treatment with prednisone

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2015-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HbA1c at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  HbA1c assessment
Change from baseline blood pressure at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  blood pressure assessments
Change from baseline cholesterol at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  cholesterol assessments
Change from baseline BMI at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  body mass index (BMI) assessments
Change from baseline weight at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  weight assessments
Change from baseline fasting glucose at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  fasting glucose assessments

SECONDARY OUTCOMES:
Change from baseline patient credential at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  Patient Credential for Diabetes Patients developed by American Pharmacists Association Foundation (APhAF)
Change from baseline depression at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  Patient Health Questionnaire 2 Question Screening (PHQ-2)
Change from baseline food security at 3, 9, 15, and 27 months | 0, 3, 9, 15, and 27 months
  Food Security Screening Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Sherr, MS, RD, CDE, Principal Investigator — American Association of Diabetes Educators
Locations (4):
- United States (4):
  - El Rio Community Health Center, Tucson, Arizona
  - Cross Trails Medical Center, Cape Girardeau, Missouri
  - Triad Adult and Pediatric Medicine, Inc., High Point, North Carolina
  - FamilyCare Health Center, Scott Depot, West Virginia